CLINICAL TRIAL: NCT07240038
Title: Evaluation of an Evidence Based, Bundled Intervention to Reduce Incidence of Ventilator-associated Pneumonia in Neonatal Units (INBERNAV-Neo)
Brief Title: Reduction of the Incidence of NAV in Neonatal Units (INBERNAV-Neo)
Acronym: INBERNAV-Neo
Status: Recruiting | Type: Observational
Sponsor: Biobizkaia Health Research Institute (Other Government)
Collaborators: Carlos III Health Institute (Other Government); Instituto de Investigacion Sanitaria La Fe (Other); European Union (Other); Hospital Universitario 12 de Octubre (Other); Hospital HM Montepríncipe (Unknown); Hospital General Universitario Gregorio Marañon (Other); Hospital Universitario La Paz (Other); Clinica Universidad de Navarra, Universidad de Navarra (Other); Hospital General Universitario de Castellón (Other); Hospital Clínico Universitario de Valencia (Other); Hospital Donostia (Other); Hospital de Basurto (Other); Complejo Hospitalario Universitario de Pontevedra (Other); Hospital Universitario de Burgos (Other); Hospital Clinico Universitario de Santiago (Other); Hospital Universitari de la Vall de Hebron (Unknown); Hospital of Navarra (Other); Hospital San Pedro de Alcantara (Other); Hospital Materno-Infantil de Canarias. Las Palmas de Gran Canaria. Spain (Unknown); Hospital Universitario Central de Asturias (Other); Hospital Universitario Marqués de Valdecilla (Other); Hospital Universitario Virgen del Rocio (Unknown); Complejo Hospitalario de Jaen (Unknown); Hospital Universitario Puerta del Mar (Other); Hospital Universitario de Jerez de la Frontera (Unknown); Hospital Materno-Infantil de Málaga (Other); Hospital General Universitario Santa Lucía (Other); Hospital Universitario Virgen de la Arrixaca (Other); Hospital Universitario La Fe (Other); Salamanca University Hospital (Other); Complexo Hospitalario Universitario de A Coruña (Other); Red Salud Materno Infantil y del Desarrollo (Other); Hospital de la Santa creu i Sant Pau - Barcelona (Other); University Hospital Virgen de las Nieves (Other); Germans Trias i Pujol Hospital (Other); Hospital del Rio Hortega (Other); Hospital Arnau de Vilanova (Other)
Responsible Party: Principal Investigator, Maria Cruz López Herrera, Lead investigator, Biobizkaia Health Research Institute
Other Study IDs: INBERNAV-Neo-21/01513; PI2024002 (Other: CEIm Euskadi)
Record Dates: First submitted 2025-06-17; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Pneumonia Ventilator Associated; Pneumonia Neonatal; Healthcare-associated Infections
Keywords: neonate; ventilator-associated pneumonia; quasi-experimental; multicenter; prevention; epidemiologic surveillance; clinical diagnosis; microbiological diagnostics; NICU; intervention; good clinical practice; patient safety
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 365 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted to participating NICUs who require mechanical ventilation
  Interventions: Behavioral: Multimodal intervention to reduce the incidence of ventilator-associated pneumonia by training the health care team in specific and general evidence-based good clinical practices.; Diagnostic Test: Technique with a blind-protected catheter

INTERVENTIONS:
Behavioral: Multimodal intervention to reduce the incidence of ventilator-associated pneumonia by training the health care team in specific and general evidence-based good clinical practices. — Bibliographical search and analysis to identify and prioritize effective and feasible interventions and procedures. Consensus among professionals for its adaptation to our Healthcare System. Areas of intervention:
  Hand hygiene: before and after patient contact and handling of respiratory equipment.
  Intubation: new and sterile ETT every intubation attempt; no contact with any non-sterile surface before insertion; avoid reintubation; ≥ two professionals.
  Suctioning: obstruction or increased respiratory secretions, never routinely. Two professional. Double suction system: one for oral cavity and one for airway, both connected to a closed suction system. Prior to ETT manipulation, patient repositioning, extubation or reintubation.
  Feeding: adjust to avoid large debris and/or distension. Positioning: lateral decubitus; head 15-30°; lateral left after feeding. Oral care: Sterile water or breast milk before intubation; every 4 h and before orogastric tube insertion. .
Diagnostic Test: Technique with a blind-protected catheter — Through the use of an invasive technique with a blind-protected catheter, the possibility of contamination and the incidence of polymicrobial etiology is reduced, resulting in a sensitive and accurate diagnosis. The method employed in this study has previously been shown to be feasible, reproducible, safe, and comparable to bronchoscopic methods for identifying VAP in children, providing sterile access to the lower respiratory tract.

SUMMARY:
The aim of this project is to achieve useful, universal and standardized definitions for the diagnosis and prevention of ventilator-associated neumonia in patients in the Neonatal Intensive Care Unit (NICU). To this end, a set of recommendations and best practice protocols have been developed in which the healthcare team of the participating units will be trained. These protocols will include evidence-based recommendations for daily practice (oral care, suctioning practices, patient positioning...) and guidelines for the diagnosis, with the goal of improving and standardizing the care that is currently carried out in each unit.

To evaluate the extent to which this intervention helps to reduce the frequency of ventilator-associated pneumonia and minimize its impact, a surveillance registry of the patient on invasive mechanical ventilation will be carried out. This registry consists of the collection of general data (sex, type of delivery, gestational age...), the drugs used during the registry (use or not of antibiotics) and the duration of the period during which the patient is under surveillance. If the patient develops pneumonia during the duration of intubation, the clinical and radiological (and in some cases microbiological) data necessary for its diagnosis and the treatment used will be collected.

The study is composed of several phases, but if we exclude the phases of formation and structure of the teams, literature review, resource preparation and data processing, the study is composed of 3 clearly differentiated phases in which patients are included. In the first phase, the coordinating team will only give the researchers of each hospital access to the forms and a brief explanation of how to fill them in, but instructing them to follow the usual diagnostic criteria. Once an established period of time has finished, the whole team belonging to the NICUs included in the project will be trained. Finally, after the training period, the teams will incorporate the preventive measures and diagnostic criteria seen in the training to their usual practice. To track behavioral changes from one phase to the next, the researchers will fill out forms to monitor the implementation of measures. Once this last phase has been completed, the results obtained will be analysed and the changes in prevention and diagnosis will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to participating NICUs who are in IMV for at least 48 hours, regardless of birth weight, gestational age or medical condition.

Exclusion Criteria:

* Patients who remain in IMV less than 48 hours.
* Decision of the healthcare professional in charge of the patient's treatment to exclude their participation at any moment due to the considerations of necessity.

Ages: 0 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients from Spanish level III and II NICUs with an average annual incidence of at least 5 neonatal patients on invasive mechanical ventilation (IMV) for ≥ 48 hours, who agree to participate and form teams to implement the best practice bundles developed to improve the care of patients on IMV. The included patients will be admitted neonates requiring IMV, regardless of birth weight or gestational age.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effect of a multimodal intervention, based on good clinical practices for the clinical management of neonates on invasive ventilatory support, on the incidence of VAP in neonates admitted to Spanish NICUs. | From the initiation of IMV until extubation plus an additional 2 days of monitoring in some cases.

SECONDARY OUTCOMES:
Systematic literature review to identify the best available scientific evidence for the unification of diagnostic criteria for VAP in neonates, and to propose evidence-based preventive measures. | An initial literature collection period of 9 months, followed by continuous updates throughout 2 years.
  The search will be conducted in major biomedical databases (PubMed, EMBASE, Cochrane Library, Scopus). The strategy will use MeSH and keywords related to VAP and neonatal populations, such as "ventilator-associated pneumonia," "VAP," "neonatal," and "mechanical ventilation." Filters will limit results to English and Spanish publications from 2015-2023, with periodic updates. Studies included will be randomized trials, cohort, case-control, reviews, and meta-analyses that assess preventive interventions or diagnostic procedures for VAP in neonates. Selected studies must describe applied methods and report quantifiable outcomes for VAP incidence or reduction. The analysis will focus on neonatal care, especially in NICUs. This approach enables synthesis of high-quality evidence, standardizes criteria, and identifies effective preventive strategies. The review will document practical interventions (hand hygiene, patient positioning, early extubation) and knowledge gaps.
Secure and user-friendly web-based registry system (Neo-NAV) for participating centers to record episodes of invasive mechanical ventilation (and VAP, if present) in neonates. | 28 months.
  This registry will collect demographic, clinical, and diagnostic data, including clinical, radiological, and microbiological criteria. Standardized forms will ensure consistency across centers, capturing variables such as coded patient ID, date of VAP diagnosis, criteria used, lab and imaging results, and treatments. The coordinating team will monitor and analyze data, communicate directly with participating centers, and prepare global reports for all investigators. This process will support comparison of diagnostic practices and assessment of inter-center variability. Data security and confidentiality will be ensured via regulatory compliance, restricted access, and audit systems. The platform will promote multicenter collaboration, enhance VAP surveillance, and improve NICU quality.
Certified and interactive online course on the Moodle platform for training healthcare professionals in standardized diagnosis and prevention of neonatal VAP. | 15 months.
  Based on the literature, training materials will be developed to unify diagnostic criteria and establish evidence-based preventive guidelines. The course will feature modules on neonatal VAP definition and epidemiology, consensus diagnostic criteria (clinical, radiological, and microbiological), and evidence-based preventive measures such as hand hygiene, ventilator care, patient positioning, and weaning. Additional topics include implementation, data recording, and quality monitoring. The platform will offer multimedia, forums, protocols, and certification assessments, with expert validation, instructional design, pilot testing, and ongoing refinement. Participants get methodological and technical support throughout the one-month course and indefinite access to materials and forums. Seven editions will be held to ensure full staff training at all participating centers.
To provide information and training on the use of telescoping catheter techniques for diagnostic purposes. | 15 months.
  In addition to unifying diagnostic criteria and implementing preventive measures, training in microbiological diagnosis using the telescoping catheter constitutes a specific component integrated into the project's training program. This technique is currently considered the most suitable for ensuring accurate diagnosis and demonstrates greater sensitivity compared to other more widely used methods. This component is addressed within the online course through a detailed video tutorial, a standardized protocol, and an infographic highlighting key concepts. Adoption of this technique in routine practice by hospitals (in cases where it was not previously implemented) will be evaluated through data reported in the Neo-NAV registry system.
. Development of a dedicated section within the Neo-NAV platform for recording preventive measures implemented against VAP in neonates at each participating hospital. | Every 4 months during a 20-month period.
  Every four months, collaborating investigators from participating centers will enter standardized data on adherence to and effectiveness of preventive bundles, including hand hygiene, ventilator circuit care, endotracheal tube management, patient positioning, among others. At the initial meeting, before the start of training, centers will register all VAP preventive measures in use and provide information on the existing protocols for intubation, extubation, and cleaning practices. In subsequent meetings, centers will update the platform with any changes implemented. This process will allow monitoring of practice modifications and their impact on recorded episodes of pneumonia.
Standardization of a definition of VAP in neonates. | 6 months.
  Diagnostic practices for VAP in neonates will be systematically documented across participating hospitals during the pre-intervention phase. This process will include recording, via the Neo-NAV platform, the application and frequency of clinical, radiological, and/or microbiological criteria routinely used for diagnosis, as well as collecting complementary information through specifically designed surveys. This will establish a baseline reference against which future interventions aimed at diagnostic standardization and improvement can be evaluated, and will also allow characterization of inter-institutional variability in diagnostic approaches and concordance among criteria applied.
Collection and analysis of antibiotic use data in the treatment of neonatal VAP. | 28 months.
  This system will record both empirical and definitive antibiotic therapies prescribed for suspected VAP, including the drug administered and treatment duration while the patient remains under invasive mechanical ventilation (IMV). In addition, all antibiotic therapies administered during IMV for infections not related to VAP will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cruz Lopez Herrera, Study Director — Biobizkaia Health Research Institute
Locations (39):
- Spain (39):
  - Hospital Universitario de A Coruña, A Coruña, A Coruña
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Complejo Hospitalario Universitario de Albacete, Albacete, Albacete
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebrón, Barcelona, Barcelona
  - Hospital Universitario de Cruces, Barakaldo, Bizkaia
  - Hospital Universitario de Basurto, Bilbao, Bizkaia
  - Hospital Universitario de Burgos (HUBU), Burgos, Burgos
  - Hospital San Pedro de Alcántara, Cáceres, Caceres
  - Hospital Universitario Puerta del Mar, Cadiz, Cadiz
  - Hospital Universitario De Jerez, Jerez de la Frontera, Cadiz
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Donostia, Donostia / San Sebastian, Gipuzkoa
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Complejo Hospitalario de Jaén, Jaén, Jaen
  - Hospital Materno Infantil de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario de León, León, Leon
  - Hospital Universitario Arnau de Vilanova, Lleida, Lleida
  - Hospital Universitario HM Monteprincipe, Boadilla del Monte, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Clínica Universidad de Navarra, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Regional Universitario de Málaga, Málaga, Malaga
  - Hospital General Universitario Santa Lucía, Cartagena, Murcia
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Murcia
  - Clínica Universidad de Navarra - Hospital, Pamplona, Navarre
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Complejo Hospitalario Universitario de Pontevedra, Pontevedra, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Clínico Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Universitario Nuestra Señora de Valme, Seville, Sevilla
  - Hospital General Universitario de Castellón, Castellon, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia
  - Hospital Universitario Río Hortega, Valladolid, Valladolid
  - Hospital Universitario Materno Infantil Miguel Servet, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Williams L. Ventilator-Associated Pneumonia Precautions for Children: What Is the Evidence? AACN Adv Crit Care. 2019 Spring;30(1):68-71. doi: 10.4037/aacnacc2019812. No abstract available. PMID 30842077
- [Background] Williams EE, Arattu Thodika FMS, Chappelow I, Chapman-Hatchett N, Dassios T, Greenough A. Diaphragmatic electromyography during a spontaneous breathing trial to predict extubation failure in preterm infants. Pediatr Res. 2022 Oct;92(4):1064-1069. doi: 10.1038/s41390-022-02085-w. Epub 2022 May 6. PMID 35523885
- [Background] WHO Guidelines on Hand Hygiene in Health Care: First Global Patient Safety Challenge Clean Care Is Safer Care. Geneva: World Health Organization; 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK144013/ PMID 23805438
- [Background] Wang L, Du KN, Zhao YL, Yu YJ, Sun L, Jiang HB. Risk Factors of Nosocomial Infection for Infants in Neonatal Intensive Care Units: A Systematic Review and Meta-Analysis. Med Sci Monit. 2019 Nov 1;25:8213-8220. doi: 10.12659/MSM.917185. PMID 31675354
- [Background] Wang HC, Liao CC, Chu SM, Lai MY, Huang HR, Chiang MC, Fu RH, Hsu JF, Tsai MH. Impacts of Multidrug-Resistant Pathogens and Inappropriate Initial Antibiotic Therapy on the Outcomes of Neonates with Ventilator-Associated Pneumonia. Antibiotics (Basel). 2020 Oct 30;9(11):760. doi: 10.3390/antibiotics9110760. PMID 33143219
- [Background] van Leuteren RW, de Waal CG, de Jongh FH, Bem RA, van Kaam AH, Hutten G. Diaphragm Activity Pre and Post Extubation in Ventilated Critically Ill Infants and Children Measured With Transcutaneous Electromyography. Pediatr Crit Care Med. 2021 Nov 1;22(11):950-959. doi: 10.1097/PCC.0000000000002828. PMID 34534162
- [Background] Tusor N, De Cunto A, Basma Y, Klein JL, Meau-Petit V. Ventilator-associated pneumonia in neonates: the role of point of care lung ultrasound. Eur J Pediatr. 2021 Jan;180(1):137-146. doi: 10.1007/s00431-020-03710-8. Epub 2020 Jun 26. PMID 32592026
- [Background] Thibeau S, Boudreaux C. Exploring the use of mothers' own milk as oral care for mechanically ventilated very low-birth-weight preterm infants. Adv Neonatal Care. 2013 Jun;13(3):190-7. doi: 10.1097/ANC.0b013e318285f8e2. PMID 23722491
- [Background] Thatrimontrichai A, Rujeerapaiboon N, Janjindamai W, Dissaneevate S, Maneenil G, Kritsaneepaiboon S, Tanaanantarak P. Outcomes and risk factors of ventilator-associated pneumonia in neonates. World J Pediatr. 2017 Aug;13(4):328-334. doi: 10.1007/s12519-017-0010-0. Epub 2017 Jan 25. PMID 28120236
- [Background] Tan B, Zhang F, Zhang X, Huang YL, Gao YS, Liu X, Li YL, Qiu JF. Risk factors for ventilator-associated pneumonia in the neonatal intensive care unit: a meta-analysis of observational studies. Eur J Pediatr. 2014 Apr;173(4):427-34. doi: 10.1007/s00431-014-2278-6. Epub 2014 Feb 13. PMID 24522325
- [Background] Ryan RM, Wilding GE, Wynn RJ, Welliver RC, Holm BA, Leach CL. Effect of enhanced ultraviolet germicidal irradiation in the heating ventilation and air conditioning system on ventilator-associated pneumonia in a neonatal intensive care unit. J Perinatol. 2011 Sep;31(9):607-14. doi: 10.1038/jp.2011.16. Epub 2011 Mar 24. PMID 21436785
- [Background] Rosenthal VD, Alvarez-Moreno C, Villamil-Gomez W, Singh S, Ramachandran B, Navoa-Ng JA, Duenas L, Yalcin AN, Ersoz G, Menco A, Arrieta P, Bran-de Casares AC, de Jesus Machuca L, Radhakrishnan K, Villanueva VD, Tolentino MC, Turhan O, Keskin S, Gumus E, Dursun O, Kaya A, Kuyucu N. Effectiveness of a multidimensional approach to reduce ventilator-associated pneumonia in pediatric intensive care units of 5 developing countries: International Nosocomial Infection Control Consortium findings. Am J Infect Control. 2012 Aug;40(6):497-501. doi: 10.1016/j.ajic.2011.08.005. Epub 2011 Nov 3. PMID 22054689
- [Background] Rosenthal VD, Al-Abdely HM, El-Kholy AA, AlKhawaja SAA, Leblebicioglu H, Mehta Y, Rai V, Hung NV, Kanj SS, Salama MF, Salgado-Yepez E, Elahi N, Morfin Otero R, Apisarnthanarak A, De Carvalho BM, Ider BE, Fisher D, Buenaflor MCSG, Petrov MM, Quesada-Mora AM, Zand F, Gurskis V, Anguseva T, Ikram A, Aguilar de Moros D, Duszynska W, Mejia N, Horhat FG, Belskiy V, Mioljevic V, Di Silvestre G, Furova K, Ramos-Ortiz GY, Gamar Elanbya MO, Satari HI, Gupta U, Dendane T, Raka L, Guanche-Garcell H, Hu B, Padgett D, Jayatilleke K, Ben Jaballah N, Apostolopoulou E, Prudencio Leon WE, Sepulveda-Chavez A, Telechea HM, Trotter A, Alvarez-Moreno C, Kushner-Davalos L; Remaining authors. International Nosocomial Infection Control Consortium report, data summary of 50 countries for 2010-2015: Device-associated module. Am J Infect Control. 2016 Dec 1;44(12):1495-1504. doi: 10.1016/j.ajic.2016.08.007. Epub 2016 Oct 11. PMID 27742143
- [Background] Raycheva R, Rangelova V, Kevorkyan A. Cost Analysis for Patients with Ventilator-Associated Pneumonia in the Neonatal Intensive Care Unit. Healthcare (Basel). 2022 May 25;10(6):980. doi: 10.3390/healthcare10060980. PMID 35742032
- [Background] Ramirez-Estrada S, Pena-Lopez Y, Vieceli T, Rello J. Ventilator-associated events: From surveillance to optimizing management. J Intensive Med. 2022 Nov 12;3(3):204-211. doi: 10.1016/j.jointm.2022.09.004. eCollection 2023 Jul 31. PMID 37533808
- [Background] Rallis D, Ben-David D, Woo K, Robinson J, Beadles D, Spyropoulos F, Christou H, Cataltepe S. Predictors of successful extubation from volume-targeted ventilation in extremely preterm neonates. J Perinatol. 2024 Feb;44(2):250-256. doi: 10.1038/s41372-023-01849-4. Epub 2023 Dec 20. PMID 38123799
- [Background] Pittet D, Hugonnet S, Harbarth S, Mourouga P, Sauvan V, Touveneau S, Perneger TV. Effectiveness of a hospital-wide programme to improve compliance with hand hygiene. Infection Control Programme. Lancet. 2000 Oct 14;356(9238):1307-12. doi: 10.1016/s0140-6736(00)02814-2. PMID 11073019
- [Background] Pinilla-Gonzalez A, Solaz-Garcia A, Parra-Llorca A, Lara-Canton I, Gimeno A, Izquierdo I, Vento M, Cernada M. Preventive bundle approach decreases the incidence of ventilator-associated pneumonia in newborn infants. J Perinatol. 2021 Jun;41(6):1467-1473. doi: 10.1038/s41372-021-01086-7. Epub 2021 May 25. PMID 34035449
- [Background] Pinilla-Gonzalez A, Lara-Canton I, Torrejon-Rodriguez L, Parra-Llorca A, Aguar M, Kuligowski J, Pineiro-Ramos JD, Sanchez-Illana A, Navarro AG, Vento M, Cernada M. Early molecular markers of ventilator-associated pneumonia in bronchoalveolar lavage in preterm infants. Pediatr Res. 2023 May;93(6):1559-1565. doi: 10.1038/s41390-022-02271-w. Epub 2022 Sep 7. PMID 36071239
- [Background] Parker LA, Weaver M, Murgas Torrazza RJ, Shuster J, Li N, Krueger C, Neu J. Effect of Gastric Residual Evaluation on Enteral Intake in Extremely Preterm Infants: A Randomized Clinical Trial. JAMA Pediatr. 2019 Jun 1;173(6):534-543. doi: 10.1001/jamapediatrics.2019.0800. PMID 31034045
- [Background] Ohnstad MO, Stensvold HJ, Pripp AH, Tvedt CR, Jelsness-Jorgensen LP, Astrup H, Eriksen BH, Klingenberg C, Mreihil K, Pedersen T, Rettedal S, Selberg TR, Solberg R, Stoen R, Ronnestad AE; Norwegian Neonatal Network. Predictors of extubation success: a population-based study of neonates below a gestational age of 26 weeks. BMJ Paediatr Open. 2022 Aug;6(1):e001542. doi: 10.1136/bmjpo-2022-001542. PMID 36053650
- [Background] Niedzwiecka T, Patton D, Walsh S, Moore Z, O'Connor T, Nugent L. What are the effects of care bundles on the incidence of ventilator-associated pneumonia in paediatric and neonatal intensive care units? A systematic review. J Spec Pediatr Nurs. 2019 Oct;24(4):e12264. doi: 10.1111/jspn.12264. Epub 2019 Jul 23. PMID 31332968
- [Background] Mohsen N, Nasef N, Ghanem M, Yeung T, Deekonda V, Ma C, Kajal D, Baczynski M, Jain A, Mohamed A. Accuracy of lung and diaphragm ultrasound in predicting successful extubation in extremely preterm infants: A prospective observational study. Pediatr Pulmonol. 2023 Feb;58(2):530-539. doi: 10.1002/ppul.26223. Epub 2022 Nov 11. PMID 36324211
- [Background] Manzoni P, De Luca D, Stronati M, Jacqz-Aigrain E, Ruffinazzi G, Luparia M, Tavella E, Boano E, Castagnola E, Mostert M, Farina D. Prevention of nosocomial infections in neonatal intensive care units. Am J Perinatol. 2013 Feb;30(2):81-8. doi: 10.1055/s-0032-1333131. Epub 2013 Jan 4. PMID 23292914
- [Background] Lin Y, Sun Z, Wang H, Liu M. The Effects of Gastrointestinal Function on the Incidence of Ventilator-associated Pneumonia in Critically Ill Patients. Open Med (Wars). 2018 Dec 6;13:556-561. doi: 10.1515/med-2018-0082. eCollection 2018. PMID 30564634
- [Background] Lambe KA, Lydon S, Madden C, Vellinga A, Hehir A, Walsh M, O'Connor P. Hand Hygiene Compliance in the ICU: A Systematic Review. Crit Care Med. 2019 Sep;47(9):1251-1257. doi: 10.1097/CCM.0000000000003868. PMID 31219838
- [Background] Klompas M, Branson R, Cawcutt K, Crist M, Eichenwald EC, Greene LR, Lee G, Maragakis LL, Powell K, Priebe GP, Speck K, Yokoe DS, Berenholtz SM. Strategies to prevent ventilator-associated pneumonia, ventilator-associated events, and nonventilator hospital-acquired pneumonia in acute-care hospitals: 2022 Update. Infect Control Hosp Epidemiol. 2022 Jun;43(6):687-713. doi: 10.1017/ice.2022.88. Epub 2022 May 20. PMID 35589091
- [Background] Jacobs Pepin B, Lesslie D, Berg W, Spaulding AB, Pokora T. ZAP-VAP: A Quality Improvement Initiative to Decrease Ventilator-Associated Pneumonia in the Neonatal Intensive Care Unit, 2012-2016. Adv Neonatal Care. 2019 Aug;19(4):253-261. doi: 10.1097/ANC.0000000000000635. PMID 31246616
- [Background] Iosifidis E, Pitsava G, Roilides E. Ventilator-associated pneumonia in neonates and children: a systematic analysis of diagnostic methods and prevention. Future Microbiol. 2018 Sep;13:1431-1446. doi: 10.2217/fmb-2018-0108. Epub 2018 Sep 26. PMID 30256161
- [Background] Hunt KA, Hunt I, Ali K, Dassios T, Greenough A. Prediction of extubation success using the diaphragmatic electromyograph results in ventilated neonates. J Perinat Med. 2020 Jul 28;48(6):609-614. doi: 10.1515/jpm-2020-0129. PMID 32598319
- [Background] Gurskis V, Asembergiene J, Kevalas R, Miciuleviciene J, Pavilonis A, Valinteliene R, Dagys A. Reduction of nosocomial infections and mortality attributable to nosocomial infections in pediatric intensive care units in Lithuania. Medicina (Kaunas). 2009;45(3):203-13. PMID 19357450
- [Background] Gupta D, Greenberg RG, Sharma A, Natarajan G, Cotten M, Thomas R, Chawla S. A predictive model for extubation readiness in extremely preterm infants. J Perinatol. 2019 Dec;39(12):1663-1669. doi: 10.1038/s41372-019-0475-x. Epub 2019 Aug 27. PMID 31455825
- [Background] Gupta A, Kapil A, Kabra SK, Lodha R, Sood S, Dhawan B, Das BK, Sreenivas V. Assessing the impact of an educational intervention on ventilator-associated pneumonia in a pediatric critical care unit. Am J Infect Control. 2014 Feb;42(2):111-5. doi: 10.1016/j.ajic.2013.09.026. PMID 24485367
- [Background] Gomez-Rios MA, Sastre JA, Lopez T, Gaszynski T. Disinfection of Reusable Laryngoscopes: A Survey about the Clinical Practice in Spain. Healthcare (Basel). 2023 Apr 13;11(8):1117. doi: 10.3390/healthcare11081117. PMID 37107952
- [Background] Gokce IK, Kutman HGK, Uras N, Canpolat FE, Dursun Y, Oguz SS. Successful Implementation of a Bundle Strategy to Prevent Ventilator-Associated Pneumonia in a Neonatal Intensive Care Unit. J Trop Pediatr. 2018 Jun 1;64(3):183-188. doi: 10.1093/tropej/fmx044. PMID 28575489
- [Background] Goerens A, Lehnick D, Buttcher M, Daetwyler K, Fontana M, Genet P, Lura M, Morgillo D, Pilgrim S, Schwendener-Scholl K, Regamey N, Neuhaus TJ, Stocker M. Neonatal Ventilator Associated Pneumonia: A Quality Improvement Initiative Focusing on Antimicrobial Stewardship. Front Pediatr. 2018 Sep 24;6:262. doi: 10.3389/fped.2018.00262. eCollection 2018. PMID 30320046
- [Background] Glowicz JB, Landon E, Sickbert-Bennett EE, Aiello AE, deKay K, Hoffmann KK, Maragakis L, Olmsted RN, Polgreen PM, Trexler PA, VanAmringe MA, Wood AR, Yokoe D, Ellingson KD. SHEA/IDSA/APIC Practice Recommendation: Strategies to prevent healthcare-associated infections through hand hygiene: 2022 Update. Infect Control Hosp Epidemiol. 2023 Mar;44(3):355-376. doi: 10.1017/ice.2022.304. Epub 2023 Feb 8. PMID 36751708
- [Background] Gauvin F, Dassa C, Chaibou M, Proulx F, Farrell CA, Lacroix J. Ventilator-associated pneumonia in intubated children: comparison of different diagnostic methods. Pediatr Crit Care Med. 2003 Oct;4(4):437-43. doi: 10.1097/01.PCC.0000090290.53959.F4. PMID 14525638
- [Background] Garland JS. Strategies to prevent ventilator-associated pneumonia in neonates. Clin Perinatol. 2010 Sep;37(3):629-43. doi: 10.1016/j.clp.2010.05.003. PMID 20813275
- [Background] Gao Y, Yin H, Wang MH, Gao YH. Accuracy of lung and diaphragm ultrasound in predicting infant weaning outcomes: a systematic review and meta-analysis. Front Pediatr. 2023 Sep 6;11:1211306. doi: 10.3389/fped.2023.1211306. eCollection 2023. PMID 37744441
- [Background] Foglia E, Meier MD, Elward A. Ventilator-associated pneumonia in neonatal and pediatric intensive care unit patients. Clin Microbiol Rev. 2007 Jul;20(3):409-25, table of contents. doi: 10.1128/CMR.00041-06. PMID 17630332
- [Background] Ezzeldin Z, Mansi Y, Gaber M, Zakaria R, Fawzy R, Mohamed MA. Nebulized hypertonic saline to prevent ventilator associated pneumonia in premature infants, a randomized trial. J Matern Fetal Neonatal Med. 2018 Nov;31(22):2947-2952. doi: 10.1080/14767058.2017.1359826. Epub 2017 Aug 8. PMID 28738709
- [Background] Esteban E, Ferrer R, Urrea M, Suarez D, Rozas L, Balaguer M, Palomeque A, Jordan I. The impact of a quality improvement intervention to reduce nosocomial infections in a PICU. Pediatr Crit Care Med. 2013 Jun;14(5):525-32. doi: 10.1097/PCC.0b013e31828a87cc. PMID 23867430
- [Background] El Amrousy D, Elgendy M, Eltomey M, Elmashad AE. Value of lung ultrasonography to predict weaning success in ventilated neonates. Pediatr Pulmonol. 2020 Sep;55(9):2452-2456. doi: 10.1002/ppul.24934. Epub 2020 Jul 8. PMID 32609928
- [Background] Sonmez Duzkaya D, Yildiz S. Effect of two different feeding methods on preventing ventilator associated pneumonia in the paediatric intensive care unit (PICU): A randomised controlled study. Aust Crit Care. 2016 Aug;29(3):139-45. doi: 10.1016/j.aucc.2015.11.001. Epub 2015 Dec 2. PMID 26652811
- [Background] Dang J, He L, Li C. Risk factors for neonatal VAP: A retrospective cohort study. Exp Biol Med (Maywood). 2023 Dec;248(23):2473-2480. doi: 10.1177/15353702231220673. Epub 2023 Dec 30. PMID 38159075
- [Background] Claassen CC, Keenan WJ. Challenging the "Culture" of the Tracheal Aspirate. Neoreviews. 2019 Mar;20(3):e145-e151. doi: 10.1542/neo.20-3-e145. PMID 31261052
- [Background] Chen YH, Lin HL, Sung YH, Hsu JF, Chu SM. Analysis of predictive parameters for extubation in very low birth weight preterm infants. Pediatr Neonatol. 2023 May;64(3):274-279. doi: 10.1016/j.pedneo.2022.08.007. Epub 2022 Nov 14. PMID 36443202
- [Background] Cernada M, Brugada M, Golombek S, Vento M. Ventilator-associated pneumonia in neonatal patients: an update. Neonatology. 2014;105(2):98-107. doi: 10.1159/000355539. Epub 2013 Nov 29. PMID 24296586
- [Background] Cernada M, Aguar M, Brugada M, Gutierrez A, Lopez JL, Castell M, Vento M. Ventilator-associated pneumonia in newborn infants diagnosed with an invasive bronchoalveolar lavage technique: a prospective observational study. Pediatr Crit Care Med. 2013 Jan;14(1):55-61. doi: 10.1097/PCC.0b013e318253ca31. PMID 22791095
- [Background] Brachio SS, Gu W, Saiman L. Next Steps for Health Care-Associated Infections in the Neonatal Intensive Care Unit. Clin Perinatol. 2023 Jun;50(2):381-397. doi: 10.1016/j.clp.2023.02.001. Epub 2023 Apr 4. PMID 37201987
- [Background] Azab SF, Sherbiny HS, Saleh SH, Elsaeed WF, Elshafiey MM, Siam AG, Arafa MA, Alghobashy AA, Bendary EA, Basset MA, Ismail SM, Akeel NE, Elsamad NA, Mokhtar WA, Gheith T. Reducing ventilator-associated pneumonia in neonatal intensive care unit using "VAP prevention Bundle": a cohort study. BMC Infect Dis. 2015 Aug 6;15:314. doi: 10.1186/s12879-015-1062-1. PMID 26246314
- [Background] Arthur N, Kaur I, Carey AJ. Evaluation of the applicability of the current CDC pediatric ventilator-associated events (PedVAE) surveillance definition in the neonatal intensive care unit population. BMC Pediatr. 2022 Apr 7;22(1):185. doi: 10.1186/s12887-022-03236-y. PMID 35392855
- [Background] Alriyami A, Kiger JR, Hooven TA. Ventilator-Associated Pneumonia in the Neonatal Intensive Care Unit. Neoreviews. 2022 Jul 1;23(7):e448-e461. doi: 10.1542/neo.23-7-e448. PMID 35773508
- [Background] Aggarwal R, Plakkal N, Bhat V. Does oropharyngeal administration of colostrum reduce morbidity and mortality in very preterm infants? A randomised parallel-group controlled trial. J Paediatr Child Health. 2021 Sep;57(9):1467-1472. doi: 10.1111/jpc.15529. Epub 2021 Apr 28. PMID 33908117
- [Background] Weber CD. Applying Adult Ventilator-associated Pneumonia Bundle Evidence to the Ventilated Neonate. Adv Neonatal Care. 2016 Jun;16(3):178-90. doi: 10.1097/ANC.0000000000000276. PMID 27195470
- [Background] Abiramalatha T, Ramaswamy VV, Thanigainathan S, Pullattayil AK, Kirubakaran R. Frequency of ventilator circuit changes to prevent ventilator-associated pneumonia in neonates and children-A systematic review and meta-analysis. Pediatr Pulmonol. 2021 Jun;56(6):1357-1365. doi: 10.1002/ppul.25345. Epub 2021 Mar 13. PMID 33713572
- See also: European Centre for Disease Prevention and Control. Hand hygiene (2015) — https://www.ecdc.europa.eu/en/publications-data/directory-guidance-prevention-and-control/core-requirements-healthcare-settings-0
- See also: Ministerio de Sanidad. Seguridad del Paciente — https://seguridaddelpaciente.sanidad.gob.es/practicasSeguras/higieneDeManos/home.htm
- See also: Organización Mundial de la Salud. Report on the burden of endemic health care-associated infection worldwide. Geneva: World Health Organization (2011) — https://iris.who.int/handle/10665/80135
- See also: Osakidetza. Estrategia de Seguridad del Paciente 2030 — https://www.osakidetza.euskadi.eus/contenidos/informacion/osk_trbg_planes_programas/es_def/adjuntos/Estrategia-de-Seguridad-del-Paciente-20-30.pdf
- See also: Pneumonia (Ventilator-associated [VAP] and non-ventilatorassociated Pneumonia [PNEU]) Event. Device-associated Module PNEU. CDC (2024) — https://www.cdc.gov/nhsn/pdfs/pscmanual/6pscvapcurrent.pdf
- See also: Ventilator-Associated Event (VAE). Device-associated Module VAE. CDC (2024) — https://www.cdc.gov/nhsn/pdfs/pscmanual/10-vae_final.pdf
- See also: World Health Organization, WHO Patient Safety. Hand hygiene technical reference manual: to be used by health-care workers, trainers and observers of hand hygiene practices (2009) — https://www.who.int/publications/i/item/9789241598606